CLINICAL TRIAL: NCT00022698
Title: A Phase II Study of Oral Xeloda (Capecitabine) in Combination With Intravenous Irinotecan for Patients With Locally Advanced and/or Metastatic Colorectal Cancer
Brief Title: Capecitabine and Irinotecan in Treating Patients With Locally Advanced, Recurrent, or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML16323
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Results first posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2005-02

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Irinotecan

ARMS (2):
- Cohort 1,Initial Regimen:(Capecitabine + Irinotecan ) (Experimental): Participants will receive capecitabine (Xeloda) 1000 mg/m^2, orally, twice daily, for 14 days (Day 2 through Day 15) every 3 weeks, along with irinotecan 125 mg/m^2 as a 90-minute intravenous (IV) infusion on Day 1 and Day 8, every 3 weeks. A total of 12 cycles of treatment will be administered. At the discretion of the investigator, participants who are responding or whose disease is stable will be permitted to continue capecitabine/irinotecan combination therapy until progressive disease is documented in the post-study treatment phase. Participants not participating in post-study treatment will be followed every 3 months until time of death, loss to follow-up, or until median survival had been reached (whichever occurred first).
  Interventions: Drug: Capecitabine; Drug: Irinotecan
- Cohort 2,Amended Regimen:(Capecitabine + Irinotecan) (Experimental): Participants will receive capecitabine 900 mg/m^2, orally, twice daily, for 14 days (Day 2 through Day 15) every 3 weeks, along with irinotecan 100 mg/m^2 as a 90-minute intravenous (IV) infusion on Day 1 and Day 8, every 3 weeks. A total of 12 cycles of treatment will be administered. At the discretion of the investigator, participants who will be responding or whose disease is stable will be permitted to continue capecitabine/irinotecan combination therapy until progressive disease is documented in the post-study treatment phase. Participants not participating in post-study treatment will be followed every 3 months until time of death, loss to follow-up, or until median survival had been reached (whichever occurred first).
  Interventions: Drug: Capecitabine; Drug: Irinotecan

INTERVENTIONS:
Drug: Capecitabine
Drug: Irinotecan

SUMMARY:
PURPOSE: Phase II trial to study the effectiveness of combining capecitabine and irinotecan in treating patients who have locally advanced, recurrent, or metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary:

* Determine the overall objective response rate in patients with locally advanced, locally recurrent, or metastatic colorectal cancer treated with capecitabine and irinotecan.

Secondary:

* Determine the time to treatment failure, time to overall response, duration of overall response, duration of overall complete response, and time to progression in patients treated with this regimen.
* Determine the 1-year survival and overall survival of patients treated with this regimen.
* Determine the toxicity and safety profile of this regimen in these patients.
* Determine the feasibility of predicting responses to this regimen by the molecular profile of tumor tissue in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive oral capecitabine twice daily on days 2-15 and irinotecan IV over 90 minutes on days 1 and 8. Treatment repeats every 3 weeks for 12 courses in the absence of disease progression or unacceptable toxicity. Patients maintaining a response or stable disease after 12 courses may continue treatment at the discretion of the investigator.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 65 patients will be accrued for this study within 9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed locally advanced, locally recurrent, or metastatic colorectal adenocarcinoma
* At least 1 measurable lesion

  * At least 10 mm by spiral CT scan
  * At least 20 mm by conventional techniques
  * Bone metastases, ascites, or pleural effusions are not considered measurable disease
* No evidence of CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 80-100%

Life expectancy:

* Not specified

Hematopoietic:

* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.25 times upper limit of normal (ULN)
* ALT and AST no greater than 2.5 times ULN (5 times ULN if liver metastases present)
* Alkaline phosphatase no greater than 2.5 times ULN (5 times ULN if liver metastases present or 10 times ULN if bone metastases present)
* No known Gilbert's disease

Renal:

* Creatinine no greater than 1.5 times ULN
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* No clinically significant cardiac disease
* No congestive heart failure
* No symptomatic coronary artery disease
* No cardiac arrhythmias uncontrolled with medication
* No myocardial infarction within the past 12 months

Gastrointestinal:

* Able to swallow tablets
* No lack of physical integrity of the upper gastrointestinal tract
* No malabsorption syndrome

Other:

* No prior unanticipated severe reaction to fluoropyrimidine therapy
* No hypersensitivity to fluorouracil
* No history of uncontrolled seizures or CNS disorders
* No psychological illness or condition that would preclude study entry
* No other malignancy within the past 5 years except curatively treated basal cell skin cancer or carcinoma in situ of the cervix
* No serious infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 12 months since prior neoadjuvant or adjuvant, active or passive immunotherapy
* No concurrent active or passive immunotherapy (e.g., 17-1A antibody) for colon cancer
* No concurrent prophylactic hematopoietic growth factors

Chemotherapy:

* At least 12 months since prior neoadjuvant or adjuvant cytotoxic chemotherapy
* No prior chemotherapy for metastatic colorectal cancer
* No prior therapy with irinotecan or capecitabine
* No other concurrent cytotoxic agents

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No prior radiotherapy to measurable lesion (newly arising lesions in a previously irradiated area allowed)
* No concurrent radiotherapy

Surgery:

* At least 4 weeks since prior major surgery and recovered
* No prior organ allograft

Other:

* At least 4 weeks since prior participation in an investigational drug study
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2001-05; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- United States (17):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - St. Louis University Hospital Cancer Center, St Louis, Missouri
  - HemOnCare, P.C., Brooklyn, New York
  - Lincoln Medical and Mental Health Center, The Bronx, New York
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Charleston Hematology-Oncology, P.A., Charleston, South Carolina
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Rockwood Clinic P.S., Spokane, Washington
  - West Virginia University Hospitals, Morgantown, West Virginia

REFERENCES:
- [Result] Meropol NJ, Gold PJ, Diasio RB, Andria M, Dhami M, Godfrey T, Kovatich AJ, Lund KA, Mitchell E, Schwarting R. Thymidine phosphorylase expression is associated with response to capecitabine plus irinotecan in patients with metastatic colorectal cancer. J Clin Oncol. 2006 Sep 1;24(25):4069-77. doi: 10.1200/JCO.2005.05.2084. PMID 16943524
- [Result] Carlini LE, Meropol NJ, Bever J, Andria ML, Hill T, Gold P, Rogatko A, Wang H, Blanchard RL. UGT1A7 and UGT1A9 polymorphisms predict response and toxicity in colorectal cancer patients treated with capecitabine/irinotecan. Clin Cancer Res. 2005 Feb 1;11(3):1226-36. PMID 15709193

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 67 participants were enrolled in the study, which was conducted from 18 May 2001 to 9 December 2004 at 18 study centers in the United States.
Pre-assignment Details: Data for participants who completed 12 cycles of the study treatment is presented.
Groups:
- Cohort 1, Initial Regimen: (Capecitabine + Irinotecan): Participants received capecitabine (Xeloda) 1000 mg/m^2, orally, twice daily, for 14 days (Day 2 through Day 15) every 3 weeks, along with irinotecan 125 mg/m^2 as a 90-minute intravenous (IV) infusion on Day 1 and Day 8, every 3 weeks. A total of 12 cycles of treatment was administered. At the discretion of the investigator, participants who were responding or whose disease was stable were permitted to continue capecitabine/irinotecan combination therapy until progressive disease was documented in the post-study treatment phase. Participants not receiving post-study treatment were followed every 3 months until time of death, loss to follow-up, or until median survival had been reached (whichever occurred first).
- Cohort 2, Amended Regimen: (Capecitabine + Irinotecan): Participants received capecitabine 900 mg/m^2, orally, twice daily, for 14 days (Day 2 through Day 15) every 3 weeks, along with irinotecan 100 mg/m^2 as a 90-minute IV infusion on Day 1 and 8, every 3 weeks. A total of 12 cycles of treatment was administered. At the discretion of the investigator, participants who were responding or whose disease was stable were permitted to continue capecitabine/irinotecan combination therapy until progressive disease was documented in the post-study treatment phase. Participants not receiving post-study treatment were followed every 3 months until time of death, loss to follow-up, or until median survival had been reached (whichever occurred first).
Period: Overall Study
Arm/Group | Cohort 1, Initial Regimen: (Capecitabine + Irinotecan) | Cohort 2, Amended Regimen: (Capecitabine + Irinotecan)
Started | 15 | 52
Completed | 7 | 17
Not Completed | 8 | 35
Not completed — Adverse Event | 5 | 9
Not completed — Death | 0 | 2
Not completed — Failure to return | 0 | 1
Not completed — Refused treatment | 0 | 2
Not completed — Insufficient therapeutic response | 2 | 14
Not completed — Administrative /other | 1 | 7

BASELINE CHARACTERISTICS:
Population: The All Patients Population included participants who received at least one dose of study drug in Cohort 1 or Cohort 2.
Groups:
- Cohort 1, Initial Regimen: (Capecitabine + Irinotecan): Participants received capecitabine 1000 mg/m^2, orally, twice daily, for 14 days (Day 2 through Day 15) every 3 weeks, along with irinotecan 125 mg/m^2 as a 90-minute IV infusion on Day 1 and Day 8, every 3 weeks. A total of 12 cycles of treatment was administered. At the discretion of the investigator, participants who were responding or whose disease was stable were permitted to continue capecitabine/irinotecan combination therapy until progressive disease was documented in the post-study treatment phase. Participants not receiving post-study treatment were followed every 3 months until time of death, loss to follow-up, or until median survival had been reached (whichever occurred first).
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Initial Regimen: (Capecitabine + Irinotecan) | Cohort 2, Amended Regimen: (Capecitabine + Irinotecan) | Total
Number analyzed (Participants) | 15 | 52 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (8.3) | 61.4 (11.1) | 61.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 21 | 30
  Male | 6 | 31 | 37

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate Based on Tumor Measurement as Per Response Evaluation Criteria In Solid Tumors Version 1.0 (RECIST 1.0)
Description: Objective Response Rate (ORR) is defined as the percentage of participants with complete response (CR) or partial response (PR) according to response evaluation criteria in solid tumors (RECIST 1.0). CR is defined as the disappearance of all target and non-target lesions and normalization of tumor marker level. PR is defined as a greater than or equal to (>/=) 30% decrease in the sum of the longest diameter (LD) of the target lesions, taking as reference the baseline sum of LD. Participants who did not have a post-baseline tumor measurement were considered non-responders in the assessment of ORR.
Time Frame: Approximately 43 Months
Population: The All Patients Population included participants who received at least one dose of study drug in Cohort 1 or Cohort 2.
Measure: Number; unit: percentage of participants
Groups:
- Cohort 1, Initial Regimen:(Capecitabine + Irinotecan): Participants received capecitabine 1000 mg/m^2, orally, twice daily, for 14 days (Day 2 through Day 15) every 3 weeks, along with irinotecan 125 mg/m^2 as a 90-minute IV infusion on Day 1 and Day 8, every 3 weeks. A total of 12 cycles of treatment was administered. At the discretion of the investigator, participants who were responding or whose disease was stable were permitted to continue capecitabine/irinotecan combination therapy until progressive disease was documented in the post-study treatment phase. Participants not receiving post-study treatment were followed every 3 months until time of death, loss to follow-up, or until median survival had been reached (whichever occurred first).
Arm/Group | Cohort 1, Initial Regimen:(Capecitabine + Irinotecan) | Cohort 2, Amended Regimen: (Capecitabine + Irinotecan)
Number analyzed (Participants) | 15 | 52
percentage of participants
  CR | 7 | 2
  PR | 40 | 42

2. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression was assessed as the time from start of treatment to the time the participant was first recorded as having disease progression or died due to causes other than disease progression. If a participant never progressed while being followed, he/she was censored at the date of the last tumor assessment or the date of the last dose if no post-baseline tumor measurement was available.
Time Frame: Approximately 43 Months
Population: The All Patients Population included participants who received at least one dose of study drug in Cohort 1 or Cohort 2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1, Initial Regimen: (Capecitabine + Irinotecan) | Cohort 2, Amended Regimen: (Capecitabine + Irinotecan)
Number analyzed (Participants) | 15 | 52
months | 6.1 [3.4 to 9.0] | 7.6 [5.8 to 8.7]

3. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was assessed as the time from start of treatment to the time the participant was withdrawn due to any of the reasons such as adverse events, progressive disease, insufficient therapeutic response, death, failure to return, or refused treatment, did not cooperate or withdrew consent.
Time Frame: Approximately 43 Months
Population: The All Patients Population included participants who received at least one dose of study drug in Cohort 1 or Cohort 2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1, Initial Regimen: (Capecitabine + Irinotecan) | Cohort 2, Amended Regimen: (Capecitabine + Irinotecan)
Number analyzed (Participants) | 15 | 52
months | 5.8 [2.4 to 9.2] | 7.3 [4.6 to 9.5]

4. Secondary Outcome: Percentage of Participants With One-year Survival
Description: Survival was measured as the time from start of treatment to the date of death or till one year whichever occurred first.
Time Frame: Up to Month 12
Population: The All Patients Population included participants who received at least one dose of study drug in Cohort 1 or Cohort 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1, Initial Regimen: (Capecitabine + Irinotecan) | Cohort 2, Amended Regimen: (Capecitabine + Irinotecan)
Number analyzed (Participants) | 15 | 52
percentage of participants | 67 [43 to 91] | 71 [58 to 83]

5. Secondary Outcome: Overall Survival
Description: Overall Survival is defined as the time from start of treatment to the date of death. Participants who did not die were censored at the last date the participant was known to be alive.
Time Frame: Approximately 43 Months
Population: The All Patients Population included participants who received at least one dose of study drug in Cohort 1 or Cohort 2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1, Initial Regimen: (Capecitabine + Irinotecan) | Cohort 2, Amended Regimen: (Capecitabine + Irinotecan)
Number analyzed (Participants) | 15 | 52
months | 22.9 [10.1 to 28.2] | 20.5 [14.9 to 30.0]

6. Secondary Outcome: Time To Objective Response
Description: The time to objective response is defined as the time from start of treatment to the date of first objective response. Participants who never responded during study were censored at the last tumor assessment or the date of last dose, whichever was later, or at the date of death if occurring prior to response.
Time Frame: Approximately 43 Months
Population: The All Patients Population included participants who received at least one dose of study drug in Cohort 1 or Cohort 2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1, Initial Regimen: (Capecitabine + Irinotecan) | Cohort 2, Amended Regimen: (Capecitabine + Irinotecan)
Number analyzed (Participants) | 15 | 52
months | 5.5 [2.7 to 8.6] | 4.3 [2.6 to 9.6]

7. Secondary Outcome: Duration of Overall Response
Description: Duration of overall response was assessed from the time that measurement criteria were first met for CR/PR (whichever is first recorded) until the first date that recurrent or progressive disease was documented. It was analyzed for responders only. Participants without observed progressive disease after an objective response were censored at the date of the last tumor assessment.
Time Frame: Approximately 43 Months
Population: The All Patients Population included participants who received at least one dose of study drug in Cohort 1 or Cohort 2. Data for participants present at the time of assessment was used for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1, Initial Regimen: (Capecitabine + Irinotecan) | Cohort 2, Amended Regimen: (Capecitabine + Irinotecan)
Number analyzed (Participants) | 7 | 23
months | 7.0 [2.6 to 9.2] | 7.7 [5.8 to 11.5]

8. Secondary Outcome: Duration of Overall Complete Response
Description: The duration of overall complete response was assessed from the time that measurement criteria were met for complete response until the first date that recurrent or progressive disease was objectively documented. Participants without observed progressive disease after an objective complete response were censored at the date of the last tumor assessment.
Time Frame: Approximately 43 Months
Population: as for outcome 7
Measure: Number; unit: months
Arm/Group | Cohort 1, Initial Regimen: (Capecitabine + Irinotecan) | Cohort 2, Amended Regimen: (Capecitabine + Irinotecan)
Number analyzed (Participants) | 1 | 1
months | 12.45 | 12.68

9. Secondary Outcome: Number of Participants With Any Adverse Events, Serious Adverse Events and Deaths
Description: An adverse event (AEs) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. A serious adverse event is defined as any event which was fatal (resulted in death), life-threatening (with immediate risk of death), resulted in a new or prolongation of a current hospitalization, resulted in persistent or significant disability or incapacity, was a congenital anomaly or birth defect, considered medically significant by the investigator, required intervention to prevent one or more of the outcomes listed above.
Time Frame: Approximately 43 Months
Population: The Safety Population consisted of all participants who received at least 1 dose of any study drug and had at least one post-baseline safety assessment. This included participants in Cohort 1 and Cohort 2.
Measure: Number; unit: Number of participants
Groups:
- Total Participants (Cohort 1 + Cohort 2): Total of all reporting groups.
Arm/Group | Cohort 1, Initial Regimen: (Capecitabine + Irinotecan) | Cohort 2, Amended Regimen: (Capecitabine + Irinotecan) | Total Participants (Cohort 1 + Cohort 2)
Number analyzed (Participants) | 15 | 52 | 67
Number of participants
  Any AEs | 15 | 52 | 67
  SAEs | 10 | 25 | 35
  Deaths During Study | 0 | 3 | 3
  Deaths During Follow-up | 13 | 23 | 36

ADVERSE EVENTS:
Time Frame: Approximately 43 Months
Description: Serious adverse events and non-serious adverse events are reported in Safety Analysis Set, which consists of all participants who received at least one dose of study medication and had a safety assessment performed post-baseline.
Arm/Group | Cohort 1, Initial Regimen: (Capecitabine + Irinotecan) | Cohort 2, Amended Regimen: (Capecitabine + Irinotecan)
Serious Adverse Events (participants affected / at risk) | 10/15 | 25/52
Other Adverse Events (participants affected / at risk) | 15/15 | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, Initial Regimen: (Capecitabine + Irinotecan) (N=15) | Cohort 2, Amended Regimen: (Capecitabine + Irinotecan) (N=52)
Diarrhoea (Gastrointestinal disorders) | 2 | 5
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 6
Constipation (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Ileitis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 3
Aortic thrombosis (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Vasoconstriction (Vascular disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, Initial Regimen: (Capecitabine + Irinotecan) (N=15) | Cohort 2, Amended Regimen: (Capecitabine + Irinotecan) (N=52)
Diarrhoea (Gastrointestinal disorders) | 13 | 45
Nausea (Gastrointestinal disorders) | 13 | 34
Vomiting (Gastrointestinal disorders) | 7 | 26
Abdominal pain (Gastrointestinal disorders) | 6 | 24
Constipation (Gastrointestinal disorders) | 5 | 17
Flatulence (Gastrointestinal disorders) | 0 | 9
Dyspepsia (Gastrointestinal disorders) | 1 | 7
Abdominal pain upper (Gastrointestinal disorders) | 0 | 6
Stomatitis (Gastrointestinal disorders) | 1 | 5
Dry mouth (Gastrointestinal disorders) | 1 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 3
Ascites (Gastrointestinal disorders) | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3
Haemorrhoids (Gastrointestinal disorders) | 0 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 3
Toothache (Gastrointestinal disorders) | 1 | 2
Abdominal hernia (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 1
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Loose stools (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 8 | 32
Oedema peripheral (General disorders) | 1 | 14
Pyrexia (General disorders) | 1 | 9
Asthenia (General disorders) | 3 | 7
Mucosal inflammation (General disorders) | 2 | 5
Chest pain (General disorders) | 0 | 3
Gait disturbance (General disorders) | 1 | 1
Discomfort (General disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 | 24
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 18
Rash (Skin and subcutaneous tissue disorders) | 2 | 12
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 13
Anorexia (Metabolism and nutrition disorders) | 2 | 13
Dehydration (Metabolism and nutrition disorders) | 2 | 11
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 6 | 18
Neutropenia (Blood and lymphatic system disorders) | 5 | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 3
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 6
Candidiasis (Infections and infestations) | 0 | 3
Nasopharyngitis (Infections and infestations) | 0 | 3
Sinusitis (Infections and infestations) | 0 | 3
Gastroenteritis viral (Infections and infestations) | 1 | 1
Herpes simplex (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 0
Nail bed infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Depression (Psychiatric disorders) | 1 | 10
Insomnia (Psychiatric disorders) | 2 | 6
Anxiety (Psychiatric disorders) | 1 | 3
Headache (Nervous system disorders) | 3 | 3
Paraesthesia (Nervous system disorders) | 0 | 4
Dysgeusia (Nervous system disorders) | 1 | 3
Dizziness (Nervous system disorders) | 3 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Weight decreased (Investigations) | 3 | 4
Blood bilirubin increased (Investigations) | 0 | 4
Weight increased (Investigations) | 1 | 2
Faecal occult blood positive (Investigations) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 3
Hypotension (Vascular disorders) | 1 | 1
Hot flush (Vascular disorders) | 1 | 1
Poor venous access (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 0
Phlebothrombosis (Vascular disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 3
Haematuria (Renal and urinary disorders) | 1 | 2
Renal failure acute (Renal and urinary disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 2
Conjunctivitis (Eye disorders) | 1 | 1
Vision blurred (Eye disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 2
Bradycardia (Cardiac disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2
Ear disorder (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.